CLINICAL TRIAL: NCT05780736
Title: Prospective Evaluation of Nivolumab in Adjuvant Esophageal Carcinoma/Gastroesophageal Junction Carcinoma: A Non-interventional Study
Brief Title: A Study to Evaluate Nivolumab in the Treatment of Early Stage Esophageal or Gastroesophageal Cancer
Acronym: PROSPECT-ESO
Status: Terminated | Type: Observational
Why Stopped: A decision was made to terminate the study due to expected timelines associated with start-up, participant enrollment, ethics committee approval and data availability from the study.
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-6KX
Record Dates: First submitted 2023-02-24; First posted 2023-03-23 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Esophageal Carcinoma; Gastroesophageal Junction Carcinoma
Keywords: Nivolumab; Adjuvant; Post Marketing; Non-interventional
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort 1

SUMMARY:
The purpose of this study is to describe the effectiveness and use of nivolumab after surgery in participants with early stage (Stage II/III) Esophageal Cancer/Gastroesophageal Junction Cancer (EC/GEJC).

ELIGIBILITY:
Inclusion criteria:

1. Must provide voluntary informed consent to participate in the study before inclusion in the study
2. Must have confirmed diagnosis of resected early stage (Stage II/III) EC or GEJC (histologically or cytologically confirmed stage)
3. Physician decision to treat the participant with adjuvant nivolumab (according to the local label as per country-specific regulations) must be made prior to and independently of participation in the study

Exclusion criteria:

1. Participation in a clinical trial of an investigational drug, concurrently or within the last 30 days (Participants who have completed their participation in an interventional trial and who are only followed-up for OS can be enrolled.)
2. Prior treatment with immuno-oncologic agents, including nivolumab, for any indication
3. Participants with a current primary diagnosis of a cancer other than EC or GEJC that requires systemic or other treatment, or has not been treated curatively (as per discretion of the investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of participants from the United States and Germany with early stage (Stage II/III) EC/GEJC who received adjuvant nivolumab after resection.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-08-23 (Actual)

PRIMARY OUTCOMES:
Disease-free Survival (DFS) | Up to 42 months, death, lost to follow-up, or study withdrawal, whichever occurs first

SECONDARY OUTCOMES:
DFS in Subgroups of Interest | Up to 42 months, death, lost to follow-up, or study withdrawal, whichever occurs first
DFS Rates in Subgroups of Interest | From baseline up to 42 months
Overall Survival (OS) | Up to 42 months, death, lost to follow-up, or study withdrawal, whichever occurs first
OS Rates | From baseline up to 42 months
Progression-free Survival (PFS) | Up to 42 months, death, lost to follow-up, or study withdrawal, whichever occurs first
PFS Rates | From baseline up to 42 months
Distant Metastasis-free Survival (DMFS) | Up to 42 months, death, lost to follow-up, or study withdrawal, whichever occurs first
DMFS Rates | From baseline up to 42 months
Treatment Patterns of Adjuvant Nivolumab | From baseline up to 42 months
Treatment Patterns of Subsequent Therapy | From baseline up to 42 months
Post-recurrence Survival | Up to Month 42, death, lost to follow-up, or study withdrawal, whichever occurs first
Time To Next Treatment | From baseline up to 42 months
OS for Participants That Received Subsequent Nivolumab Treatment | Up to 42 months, death, lost to follow-up, or study withdrawal, whichever occurs first
OS Rates for Participants That Received Subsequent Nivolumab Treatment | From baseline up to 42 months
PFS for Participants That Received Subsequent Nivolumab Treatment | Up to 42 months, death, lost to follow-up, or study withdrawal, whichever occurs first
PFS Rates for Participants That Received Subsequent Nivolumab Treatment | From baseline up to 42 months
Overall Response Rate for Participants That Received Subsequent Nivolumab Treatment | From baseline up to 42 months
Time to Disease Recurrence | From baseline up to 42 months
Type of Disease Recurrence | From baseline up to 42 months
Participant Sociodemographics | From baseline up to 42 months
Number of Participants with Adverse Events | From baseline up to 42 months
Number of Participants with Serious Adverse Events Related to Nivolumab Treatment | From baseline up to 42 months
Disease stage at initial diagnosis | From baseline up to 42 months
  Esophageal Cancer/Gastroesophageal Junction Cancer (EC/GEJC) stage (i.e., I, II or III) and stage using Tumor, node, and metastasis (TNM) system
Eastern Cooperative Oncology Group (ECOG) performance status | From baseline up to 42 months
  0: Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work on a light or sedentary nature
  2. Ambulatory and capable of all self-care but unable to carry out work activities. Up and about more than 50% of waking hours
  3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair
  5. Dead
Tumor location at initial diagnosis | From baseline up to 42 months
  EC (upper, middle, lower area of the esophagus) or GEJC (Siewert type I, II or III, if available)
Tumor histology at initial diagnosis | From baseline up to 42 months
  Squamous Cell Carcinoma (SSC) or adenocarcinoma
Pathologic lymph node status | From baseline up to 42 months
  ypN0, ypN1, ypN2, ypN3, unknown
Pathologic tumor status | From baseline up to 42 months
  ypT0, ypT1, ypT2, ypT3, ypT4, unknown
Tumor cell PD-L1 expression (≥1% vs. <1% vs. indeterminate/non-evaluable) | From baseline up to 42 months
  Tumor cell PD-L1 expression levels and cells assessed. This will be used to group PD-L1 expression into ≥1%, <1%, or Indeterminate/non-evaluable and to derive the combined positive score (CPS) score which is defined as PD-L1 positive tumor cells + PD-L1 positive mononuclear inflammatory cells)/Total tumor cells) × 100
Type of recurrence | From baseline up to 42 months
  local/regional vs. distant
Serum levels of nuclear protein Ki67 | From baseline up to 42 months
Number of participants with metastasis | From baseline up to 42 months
Sites of metastases | From baseline up to 42 months
  Lung, brain, liver, peritoneum, bone, lymph nodes, other
Comorbidities | From baseline up to 42 months
  Diagnosis date and name of diagnosis, grouped using the National Cancer Institute (NCI) Comorbidity Index.
Concomitant treatments | From baseline up to 42 months
  Type of treatment or therapies receive in parallel of nivolumab treatment and details (e.g., medications, radiotherapy, chemotherapy, systemic therapy, or surgical treatment)
Concurrent medical conditions | From baseline up to 42 months
Prior treatments for EC/GEJC | From baseline up to 42 months
  Type of therapies received prior to initiation of nivolumab treatment (e.g., radiotherapy, chemotherapy, targeted therapy, systemic treatment, platinum-based therapy) and details (if applicable, e.g., regimens, dosing
Participant Treatment History | From baseline up to 42 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (24):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Pacific Central Coast Health Centers - San Luis Obispo Oncology and Hematology Health Center, San Luis Obispo, California
  - Mission Cancer Center, Santa Maria, California
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - UPMC Hillman Cancer Center, Westwood, Kansas
  - University Of Louisville, Louisville, Kentucky
  - Weill Cornell Medical College, New York, New York
  - Local Institution - 0009, Dallas, Texas
  - William Beaumont Army Medical Center, Fort Bliss, Texas
  - The University Of Texas, Houston, Texas
  - Baylor Scott and White Health, Temple, Texas
- Germany (13):
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Klinikum Munchen-Bogenhausen, München, Bavaria
  - Klinikum Kassel, Kassel, Hesse
  - Onkologische Schwerpunktpraxis Dres. Ingo Zander und Eyck von der Heyde, Hanover, Lower Saxony
  - Alexianer, Maria-Hilf-Krankenhaus, Essen, North Rhine-Westphalia
  - Oncologianova GmbH, Recklinghausen, North Rhine-Westphalia
  - Local Institution - 0006, Mainz, Rhineland-Palatinate
  - Universitätsklinikum Bonn, Bonn, Saarland
  - Local Institution - 0033, Homburg, Saarland
  - CaritasKlinikum Saarbruecken., Saarbrücken, Saarland
  - Klinikum Chemnitz Ggmbh, Chemnitz, Saxony
  - BAG Freiberg-Richter, Jacobash, Illmer, Wolf, Dresden, Saxony
  - Universitätsklinik Magdeburg, Magdeburg, Saxony-Anhalt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html